CLINICAL TRIAL: NCT05334628
Title: The Effect of Erector Spinae Plane Block on Intraoperative Hemodynamics in Video-Assisted Thoracoscopic Surgery
Brief Title: The Effect of ESPB on Intraoperative Hemodynamics in VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nilgün Zengin, Principal İnvestigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-22-2536
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Video-Assisted Thoracoscopic Surgery; Erector Spinae Plane Block; Mean Arterial Pressure; Heart Rate

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative Erector Spinae Plane Block (Active Comparator): In the preoperative period, under general anesthesia, after the linear ultrasound (US) probe will be placed 2-3 cm lateral to the T5 spinous process, 30 ml of 0.25% bupivacaine hydrochloride will be injected into the interfacial space below the erector spinae muscle, above the transverse process.
  Interventions: Procedure: Preoperative Erector spinae plane block
- Postperative Erector Spinae Plane Block (Active Comparator): In the postoperative period, under general anesthesia, after the linear ultrasound (US) probe will be placed 2-3 cm lateral to the T5 spinous process, 30 ml of 0.25% bupivacaine hydrochloride will be injected into the interfacial space below the erector spinae muscle, above the transverse process.
  Interventions: Procedure: Postperative Erector spinae plane block

INTERVENTIONS:
Procedure: Preoperative Erector spinae plane block — Erector spinae plane block will be performed unilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, and when the patient is placed in the lateral decubitus position.
  Arms: Preoperative Erector Spinae Plane Block
Procedure: Postperative Erector spinae plane block — Erector spinae plane block will be performed unilaterally, under US guidance, after the surgical operation, under general anesthesia, and when the patient is placed in the lateral decubitus position.
  Arms: Postperative Erector Spinae Plane Block

SUMMARY:
Video-assisted thoracic surgery (VATS) is frequently applied in thoracic surgery operations. VATS has become the standard procedure in minor and major lung surgeries. In recent years, regional anesthesia techniques have also been frequently applied to patients for pain relief. Thoracic paravertebral block (TPVB), erector spinae plane block (ESPB), and serratus anterior plane block (SAPB) are also among the regional anesthesia techniques frequently used in thoracic surgery.

General anesthesia (GA) is the main method of anesthesia for thoracic surgery. However, GA can only inhibit the projection system of the cortical limbic system or hypothalamic cortex. GA cannot completely block the transmission of peripheral noxious stimulus to the central nervous system and cannot effectively inhibit the intraoperative stress response. With the addition of peripheral blocks such as TPVB, ESPB, and SAPB, more stable hemodynamics is expected by providing preemptive analgesia in patients. As a result of all these; In this study, we aimed to compare the intraoperative hemodynamic changes of patients who underwent preoperative ESPB in patients who will undergo VATS resection under GA with those who underwent postoperative ESPB.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* American Society of Anesthesiologists physical status I-II-III
* Body mass index between 18-40 kg/m2
* Patients undergoing elective video assisted thoracoscopic surgery

Exclusion Criteria:

* Advanced cancer
* History of chronic analgesic therapy
* History of local anesthetic allergy
* Infection in the intervention area
* Patients with bleeding disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | Perioperative period
  Mean arterial pressure values will be recorded before anesthesia, before surgical incision, after surgical incision at 5th, 30th, 60th, 90th, 120th minutes, and after general anesthesia.
Heart rate | Perioperative period
  Heart rate values will be recorded before anesthesia, before surgical incision, after surgical incision at 5th, 30th, 60th, 90th, 120th minutes, and after general anesthesia.

SECONDARY OUTCOMES:
Pain scores | First 24 hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at the 1st, 2nd, 4th, 12th, and 24th hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Zengin, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara City Hospital, Çankaya, Ankara
  - Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara

IPD SHARING:
Plan to Share IPD: No